CLINICAL TRIAL: NCT04975048
Title: SREBF1 Polymorphism and Egg Yolk on Cardiovascular Disease Risk in Healthy Young Adults: a Randomised, Two-period, Single Blinded, Crossover Trial
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding for secondary outcomes in fecal microbiome is not solved
Sponsor: Shandong University (Other)
Collaborators: Chinese Nutrition Society (Unknown); Fudan University (Other)
Responsible Party: Principal Investigator, Shixiu Zhang, Principal Investigator, Shandong University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CNS-W2018A44
Record Dates: First submitted 2021-06-30; First posted 2021-07-23 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-05

CONDITIONS: Healthy; GEN1 Gene Mutation
Keywords: Gene-by-Diet Interaction; Egg Yolk; Sterol Regulatory Element Binding Protein 1 Gene; HDL-C; LDL-C/HDL-C
MeSH Terms: interventions — Egg Yolk

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Masking was applied for those who collected blood samples, physical examination data, and assessed laboratory outcomes. People who were masked did not participate in the routine management meetings of the trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A was consisted of 16 rs2236513/rs2297508/rs4925119 C/G/G carriers and 16 AA/CC/AA homozygotes. And it was first assigned egg yolk intervention during intervention period 1, and then macronutrient equivalent control during intervention period 2
  Interventions: Dietary Supplement: Egg yolks; Dietary Supplement: Macronutrients equivalent control
- Group B (Other): Group B was also consisted of 16 rs2236513/rs2297508/rs4925119 C/G/G carriers and 16 AA/CC/AA homozygotes. It was first assigned macronutrient equivalent control during intervention period 1, and then egg yolk during intervention period 2
  Interventions: Dietary Supplement: Egg yolks; Dietary Supplement: Macronutrients equivalent control

INTERVENTIONS:
Dietary Supplement: Egg yolks — Two egg yolks/day was designed for the study. However, uneven egg sizes during period 1 made the intervention unable to achieve the protocol's recommended cholesterol intake level, and the intervention was modified in period 2 to be 0.8 g egg yolk/day/kg body weight. This dosage was calculated by dividing the 35 g egg yolk with the lightest weight among the volunteers, which was 45 kg. This provides a more consistent cholesterol intake between persons as the egg yolk dosage is standardized for persons with different weights.
Dietary Supplement: Macronutrients equivalent control — The macronutrients equivalent control group was served 42 g egg white cooked with 10 g olive oil, designed to best imitate the energy and macronutrients of 35 g egg yolk (energy 119 kcal, protein 5 g, fat 10 g, carbohydrate 1 g) since the average weight of two large egg yolk was presumed to be 35 g. As an egg yolk dose of 0.8 g egg yolk per kg body weight per day was served during the intervention period 2, the macronutrients equivalent control was likewise adjusted as follow: subjects who weighed less than 55 kg were served 51 g egg white cooked with 12 g olive oil, which is equivalent to 40 g egg yolk; those who weighed from 55 kg to 65 kg were served 61 g egg white cooked with 14 g olive oil, which is equivalent to 48 g egg yolk; and those who weighed more than 65 kg were served 71 g egg white cooked with 17 g olive oil, which is equivalent to 56 g egg yolk.

SUMMARY:
Our previous analysis showed that sterol regulatory element binding protein gene (SREBF1) rs2236513/rs2297508/rs4925119 polymorphism modulated the relation between dietary cholesterol and serum low density lipoprotein cholesterol /serum total cholesterol. This study aims to confirm and extend this finding by characterizing the effects of cholesterol from egg yolks on lipid profiles in healthy young adults with different SREBF1 genetic makeup. 32 SREBF1 C/G/G minor allele carriers at rs2236513/rs2297508/rs4925119 and 32 SREBF1 AA/CC/AA major homozygotes at rs2236513/rs2297508/rs4925119 were enrolled to test their response to egg yolks.

ELIGIBILITY:
Inclusion Criteria:

* SREBF1 C/G/G minor allele carriers and AA/CC/AA major homozygotes at rs2236513/rs2297508/rs4925119, age 18-25 years, body mass index (BMI) 18~23.9 kg/m2 , blood pressure within normal ranges (Systolic blood pressure < 140mmHg, diastolic blood pressure < 90mmHg), lipid profiles within normal ranges according to test kit instructions (fasting serum triglycerides < 1.7mmol/L, fasting serum total cholesterol < 5.2 mmol/L, fasting serum low density lipoprotein cholesterol (LDL-C) < 3.12 mmol/L, fasting serum high density lipoprotein cholesterol (HDL-C) >1.04 mmol/L ), liver and kidney functions within normal ranges according to test kit instructions (alanine aminotransferase (ALT) 9~50 U/L for male, 7~40 U/L for female; aspartate transaminase (AST) 15~40 U/L for male, 13~35 U/L for female; creatinine 62~115 μmol/L for male, 53~97 μmol/L for female; blood urea nitrogen (BUN), 1.43~7.14 mmol/L), both parents are Chinese Han nationality, willing to eat two or more eggs, and willing to maintain "Three Low Diet" except when they were given egg yolks during the study.

Exclusion Criteria:

* History of diabetes, cancer, stroke, heart disease or any other known diseases, allergic to eggs, or having habits such as drinking or smoking.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2020-01-12 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes in serum lipids | Week 0, week 4, week 8, week 16
  Serum lipids including serum total cholesterol, LDL-C, HDL-C and LDL-C/HDL-C, triglycerides

CONTACTS AND LOCATIONS:
Overall Officials: Shixiu Zhang, Ph. D., Study Chair — Shandong University
Locations (1):
- Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol
Time Frame: All IPD that underlie results in a publication will be shared as claimed by the journal that the publication is published.
Access Criteria: Can access data by contacting Shixiu Zhang.